CLINICAL TRIAL: NCT03121625
Title: CAR-T Therapy in Relapsed or Refractory Haematopoietic and Lymphoid Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016040
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous CAR-T cells (Experimental): Patients will be be treated with autologous CAR-T cells.
  Interventions: Biological: Autologous CAR-T

INTERVENTIONS:
Biological: Autologous CAR-T — Patients will be drawn 50-100 ml blood to obtain enough peripheral blood mononuclear cells (PBMC) for CAR-T manufacturing. The T cells will be purified from the PBMC, transduced with CAR lentiviral vector, expanded in vitro and then frozen for future administration. Chemotherapy will then be given. Following tumor burden reassessment, CAR-T cells will be infused.

SUMMARY:
This is an open, single-arm, phase I clinical study to evaluate efficacy and safety of chimeric antigen receptor T cell immunotherapy (CAR-T) in the treatment of hematopoietic and lymphoid malignancies. A total of 30 patients are planned to be enrolled over a period of 2 years.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells targeted against CD19 have demonstrated unprecedented successes in treating patients with hematopoietic and lymphoid malignancies. Besides CD19, many other molecules such as CD22, CD30, CD7, BCMA, CD123, etc. may be potential in developing the corresponding CAR-T cells to treat patients whose tumors expressing those markers. Investigators have developed a high efficient platform for constructing different CARs and preclinical studies have demonstrated effective killing of corresponding target cells. In this study, investigators will evaluate their safety and efficacy in patients with different types of hematopoietic and lymphoid malignancies. The primary goal is safety assessment including cytokine storm response and any other adverse effects. In addition, tumor targeting and disease status after treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1.The treat history meeting the following criteria:

1. Recurrence of lymphoma patients with imaging (CT/MRI/PET-CT) detection and pathological diagnosis, or recurrence including bone marrow morphology relapse and the MRD recurrence of myeloma patients or leukemia patients, after chemotherapy or stem cell transplantation;
2. Can't get complete remission (including MRD positive) after more than twice repeated chemotherapy of incipient lymphoma, myeloma or leukemia patients;
3. One or twice chemotherapy cannot get remission again (including MRD positive), but not suitable for chemotherapy of incipient lymphoma, myeloma or leukemia patients.

2. There is a measurable lesions before treatment at least; 3. ECOG score≤2; 4. To be aged 1 to 70 years; 5. More than a month lifetime from the consent signing date

Exclusion Criteria:

1. Serious cardiac insufficiency, left ventricular ejection fraction<50;
2. Has a history of severe pulmonary function damaging;
3. Merging other malignant tumor;
4. Merging uncontrolled infection;
5. Merging the metabolic diseases (except diabetes);
6. Merging severe autoimmune diseases or immunodeficiency disease;
7. patients with active hepatitis B or hepatitis C;
8. patients with HIV infection;
9. Has a history of serious allergies on Biological products (including antibiotics);
10. Happened in 3 ~ 4 acute GvHD after allogeneic hematopoietic stem cell transplantation on recurring patients
11. Pregnancy or lactation women;
12. Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluation.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12-26 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Tumor load | Up to 24 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis.

SECONDARY OUTCOMES:
CAR T cell persistence | Up to 24 months]
  CAR T cell persistence will be quantified with flow cytometry and qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Lihong Liu, PhD & MD, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Hematology Department, Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided